CLINICAL TRIAL: NCT01061554
Title: Correlation Between Level of Polyunsaturated Fatty Acid EPA and DHA in Blood After Digestion of ProBios Omega-3 Concordix™ Compared With Omega-3 Soft Capsules - a Pilot
Brief Title: Bioavailability Study of Long Chain Omega-3 Fatty Acids From a Gastric Stable Emulsion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ayanda AS (Industry)
Responsible Party: Tore Seternes, Ayanda AS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AYANDA-CC-01
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2009-04

CONDITIONS: Healthy
Keywords: Bioavailability; Eicosapentaenoic acid; Docosahexaenoic acid; Soft gel capsules; Gastric stable emulsion; Omega-3; Tri-glycerides; Marine phospholipids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gastric stable emulsion (Experimental): A gastric stable emulsion vehicle for administration of tri-glyceride based omega-3 oils
  Interventions: Dietary Supplement: Omega-3 oils from tri-glycerides
- Soft gel capsule (TG) (Active Comparator): Soft gel capsule for administration of tri-glyceride based omega-3 oils
  Interventions: Dietary Supplement: Omega-3 oils from tri-glycerides
- Soft gel capsules (MPL) (Active Comparator): Soft gel capsule for administration of marine phospholipids based omega-3 oils
  Interventions: Dietary Supplement: Omega-3 oils from marine phospholipids

INTERVENTIONS:
Dietary Supplement: Omega-3 oils from tri-glycerides — Single-dose administration of approximately 5 grams of omega-3 oils from triglycerides
  Arms: Gastric stable emulsion; Soft gel capsule (TG)
Dietary Supplement: Omega-3 oils from marine phospholipids — Single-dose administration of approximately 5 grams of omega-3 oils from marine phospholipids
  Arms: Soft gel capsules (MPL)

SUMMARY:
The purpose of this study is to compare the short term absorption of EPA and DHA from triglycerides (TG) released from normal soft gel capsules and from the new patent pending vehicle providing a gastric stable emulsion.

DETAILED DESCRIPTION:
The present study comprises the design of as well as the effect of pre-emulsification of ω-3 fatty acids on the bioavailability of docosahexaenoic acid and eicosapentaenoic acid. In-vitro studies have shown that long-term steric stabilization of an o/w-emulsion is obtained by arresting the oil droplets in a gelatin continuous gel matrix. The emulsion was also stable upon dissolution of the gel matrix at physiological conditions in-vitro and is hence referred to as a gastric stable emulsion (GSE).

In the bioavailability study, healthy young students were recruited and presented two different single-dose treatments of fish oil containing 5 grams of ω-3 fatty acids; one group receiving the fatty acids in traditional soft gel capsules, whereas the other group received the fatty acids using the GSE technology. Time resolved (2 - 26 hours) blood plasma analysis after intake of this single dose ω-3 fatty acids revealed significantly increased AUC0-26h and Cmax of EPA and EPA + DHA when administered as GSE compared to traditional soft gel capsules.

ELIGIBILITY:
Inclusion Criteria:

* Student at Nord-Trondelag University College
* Healthy (no known condition)
* Males and females aged 19 to 29 years

Exclusion Criteria:

* Fish allergies
* Ongoing consumption of omega-3 fatty acids
* Subjects receiving anticoagulation or non-steroid anti-inflammatory treatment
* Subjects with a known metabolic syndrome; diabetes, hypercholesterol, hypertension, obesity

Ages: 19 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The incremental (change from baseline) area under the blood plasma concentration curve of eicosapentaenoic acid (EPA) | 26 hours (blood samples taken at baseline and 2, 3, 4, 6, 8 and 26 hours after treatment administration)
The incremental (change from baseline) area under the blood plasma concentration curve of docosahexaenoic acid (DHA) | 26 hours (blood samples taken at baseline and 2, 3, 4, 6, 8 and 26 hours after treatment administration)
The incremental (change from baseline) area under the blood plasma concentration curve of Vitamin E | 26 hours (blood samples taken at baseline and 2, 3, 4, 6, 8 and 26 hours after treatment administration)

SECONDARY OUTCOMES:
The maximal incremental blood plasma concentration of EPA | 26 hours (blood samples taken at baseline and 2, 3, 4, 6, 8 and 26 hours after treatment administration)
The maximal incremental blood plasma concentration of DHA | 26 hours (blood samples taken at baseline and 2, 3, 4, 6, 8 and 26 hours after treatment administration)
The maximal incremental blood plasma concentration of Vitamin E | 26 hours (blood samples taken at baseline and 2, 3, 4, 6, 8 and 26 hours after treatment administration)
The time passed since administration at which the incremental plasma concentration maximum occurs for EPA | 26 hours (blood samples taken at baseline and 2, 3, 4, 6, 8 and 26 hours after treatment administration)
The time passed since administration at which the incremental plasma concentration maximum occurs for DHA | 26 hours (blood samples taken at baseline and 2, 3, 4, 6, 8 and 26 hours after treatment administration)
The time passed since administration at which the incremental plasma concentration maximum occurs for Vitamin E | 26 hours (blood samples taken at baseline and 2, 3, 4, 6, 8 and 26 hours after treatment administration)

CONTACTS AND LOCATIONS:
Locations (1):
- Nord-Trøndelag University College, Namsos, Nord-Trøndelag, Norway

REFERENCES:
- [Background] Armand M, Borel P, Dubois C, Senft M, Peyrot J, Salducci J, Lafont H, Lairon D. Characterization of emulsions and lipolysis of dietary lipids in the human stomach. Am J Physiol. 1994 Mar;266(3 Pt 1):G372-81. doi: 10.1152/ajpgi.1994.266.3.G372. PMID 8166277
- [Background] Armand M, Borel P, Pasquier B, Dubois C, Senft M, Andre M, Peyrot J, Salducci J, Lairon D. Physicochemical characteristics of emulsions during fat digestion in human stomach and duodenum. Am J Physiol. 1996 Jul;271(1 Pt 1):G172-83. doi: 10.1152/ajpgi.1996.271.1.G172. PMID 8760121
- [Background] Armand M, Pasquier B, Andre M, Borel P, Senft M, Peyrot J, Salducci J, Portugal H, Jaussan V, Lairon D. Digestion and absorption of 2 fat emulsions with different droplet sizes in the human digestive tract. Am J Clin Nutr. 1999 Dec;70(6):1096-106. doi: 10.1093/ajcn/70.6.1096. PMID 10584056
- [Background] Arterburn LM, Hall EB, Oken H. Distribution, interconversion, and dose response of n-3 fatty acids in humans. Am J Clin Nutr. 2006 Jun;83(6 Suppl):1467S-1476S. doi: 10.1093/ajcn/83.6.1467S. PMID 16841856
- [Background] Arterburn LM, Oken HA, Hoffman JP, Bailey-Hall E, Chung G, Rom D, Hamersley J, McCarthy D. Bioequivalence of Docosahexaenoic acid from different algal oils in capsules and in a DHA-fortified food. Lipids. 2007 Nov;42(11):1011-24. doi: 10.1007/s11745-007-3098-5. Epub 2007 Aug 23. PMID 17713804
- [Background] Borel P, Pasquier B, Armand M, Tyssandier V, Grolier P, Alexandre-Gouabau MC, Andre M, Senft M, Peyrot J, Jaussan V, Lairon D, Azais-Braesco V. Processing of vitamin A and E in the human gastrointestinal tract. Am J Physiol Gastrointest Liver Physiol. 2001 Jan;280(1):G95-G103. doi: 10.1152/ajpgi.2001.280.1.G95. PMID 11123202
- [Background] Bucher HC, Hengstler P, Schindler C, Meier G. N-3 polyunsaturated fatty acids in coronary heart disease: a meta-analysis of randomized controlled trials. Am J Med. 2002 Mar;112(4):298-304. doi: 10.1016/s0002-9343(01)01114-7. PMID 11893369
- [Background] Cao J, Schwichtenberg KA, Hanson NQ, Tsai MY. Incorporation and clearance of omega-3 fatty acids in erythrocyte membranes and plasma phospholipids. Clin Chem. 2006 Dec;52(12):2265-72. doi: 10.1373/clinchem.2006.072322. Epub 2006 Oct 19. PMID 17053155
- [Background] Elvevoll EO, Barstad H, Breimo ES, Brox J, Eilertsen KE, Lund T, Olsen JO, Osterud B. Enhanced incorporation of n-3 fatty acids from fish compared with fish oils. Lipids. 2006 Dec;41(12):1109-14. doi: 10.1007/s11745-006-5060-3. PMID 17269556
- [Background] Elvevoll EO, Eilertsen KE, Brox J, Dragnes BT, Falkenberg P, Olsen JO, Kirkhus B, Lamglait A, Osterud B. Seafood diets: hypolipidemic and antiatherogenic effects of taurine and n-3 fatty acids. Atherosclerosis. 2008 Oct;200(2):396-402. doi: 10.1016/j.atherosclerosis.2007.12.021. Epub 2008 Feb 1. PMID 18242615
- [Background] Garaiova I, Guschina IA, Plummer SF, Tang J, Wang D, Plummer NT. A randomised cross-over trial in healthy adults indicating improved absorption of omega-3 fatty acids by pre-emulsification. Nutr J. 2007 Jan 25;6:4. doi: 10.1186/1475-2891-6-4. PMID 17254329
- [Background] Grimsgaard S, Bonaa KH, Hansen JB, Myhre ES. Effects of highly purified eicosapentaenoic acid and docosahexaenoic acid on hemodynamics in humans. Am J Clin Nutr. 1998 Jul;68(1):52-9. doi: 10.1093/ajcn/68.1.52. PMID 9665096
- [Background] Harris WS. Omega-3 fatty acids and cardiovascular disease: a case for omega-3 index as a new risk factor. Pharmacol Res. 2007 Mar;55(3):217-23. doi: 10.1016/j.phrs.2007.01.013. Epub 2007 Jan 25. PMID 17324586
- [Background] Iso H, Kobayashi M, Ishihara J, Sasaki S, Okada K, Kita Y, Kokubo Y, Tsugane S; JPHC Study Group. Intake of fish and n3 fatty acids and risk of coronary heart disease among Japanese: the Japan Public Health Center-Based (JPHC) Study Cohort I. Circulation. 2006 Jan 17;113(2):195-202. doi: 10.1161/CIRCULATIONAHA.105.581355. Epub 2006 Jan 9. PMID 16401768
- [Background] Hsu, J. C. (1992). The Factor Analytic Approach to Simultaneous Inference in the General Linear Model. Journal of Computational and Graphical Statistics, 1(2), 151-168.
- [Background] Krokan HE, Bjerve KS, Mork E. The enteral bioavailability of eicosapentaenoic acid and docosahexaenoic acid is as good from ethyl esters as from glyceryl esters in spite of lower hydrolytic rates by pancreatic lipase in vitro. Biochim Biophys Acta. 1993 May 20;1168(1):59-67. doi: 10.1016/0005-2760(93)90266-c. PMID 8504143
- [Background] Liu ZX, Artmann C. Relative bioavailability comparison of different coenzyme Q10 formulations with a novel delivery system. Altern Ther Health Med. 2009 Mar-Apr;15(2):42-6. PMID 19284181
- [Background] London B, Albert C, Anderson ME, Giles WR, Van Wagoner DR, Balk E, Billman GE, Chung M, Lands W, Leaf A, McAnulty J, Martens JR, Costello RB, Lathrop DA. Omega-3 fatty acids and cardiac arrhythmias: prior studies and recommendations for future research: a report from the National Heart, Lung, and Blood Institute and Office Of Dietary Supplements Omega-3 Fatty Acids and their Role in Cardiac Arrhythmogenesis Workshop. Circulation. 2007 Sep 4;116(10):e320-35. doi: 10.1161/CIRCULATIONAHA.107.712984. No abstract available. PMID 17768297
- [Background] Lund EK, Harvey LJ, Ladha S, Clark DC, Johnson IT. Effects of dietary fish oil supplementation on the phospholipid composition and fluidity of cell membranes from human volunteers. Ann Nutr Metab. 1999;43(5):290-300. doi: 10.1159/000012797. PMID 10749029
- [Background] Marangoni F, Angeli MT, Colli S, Eligini S, Tremoli E, Sirtori CR, Galli C. Changes of n-3 and n-6 fatty acids in plasma and circulating cells of normal subjects, after prolonged administration of 20:5 (EPA) and 22:6 (DHA) ethyl esters and prolonged washout. Biochim Biophys Acta. 1993 Dec 2;1210(1):55-62. doi: 10.1016/0005-2760(93)90049-f. PMID 8257719
- [Background] Marchioli R, Barzi F, Bomba E, Chieffo C, Di Gregorio D, Di Mascio R, Franzosi MG, Geraci E, Levantesi G, Maggioni AP, Mantini L, Marfisi RM, Mastrogiuseppe G, Mininni N, Nicolosi GL, Santini M, Schweiger C, Tavazzi L, Tognoni G, Tucci C, Valagussa F; GISSI-Prevenzione Investigators. Early protection against sudden death by n-3 polyunsaturated fatty acids after myocardial infarction: time-course analysis of the results of the Gruppo Italiano per lo Studio della Sopravvivenza nell'Infarto Miocardico (GISSI)-Prevenzione. Circulation. 2002 Apr 23;105(16):1897-903. doi: 10.1161/01.cir.0000014682.14181.f2. PMID 11997274
- [Background] Marsen TA, Pollok M, Oette K, Baldamus CA. Pharmacokinetics of omega-3-fatty acids during ingestion of fish oil preparations. Prostaglandins Leukot Essent Fatty Acids. 1992 Jul;46(3):191-6. doi: 10.1016/0952-3278(92)90069-u. PMID 1387231
- [Background] McDowell EM, Trump BF. Histologic fixatives suitable for diagnostic light and electron microscopy. Arch Pathol Lab Med. 1976 Aug;100(8):405-14. PMID 60092
- [Background] Nestel P, Shige H, Pomeroy S, Cehun M, Abbey M, Raederstorff D. The n-3 fatty acids eicosapentaenoic acid and docosahexaenoic acid increase systemic arterial compliance in humans. Am J Clin Nutr. 2002 Aug;76(2):326-30. doi: 10.1093/ajcn/76.2.326. PMID 12145002
- [Background] Obeidat WM. Recent patents review in microencapsulation of pharmaceuticals using the emulsion solvent removal methods. Recent Pat Drug Deliv Formul. 2009 Nov;3(3):178-92. doi: 10.2174/187221109789105612. PMID 19925442
- [Background] Radaelli A, Cazzaniga M, Viola A, Balestri G, Janetti MB, Signorini MG, Castiglioni P, Azzellino A, Mancia G, Ferrari AU. Enhanced baroreceptor control of the cardiovascular system by polyunsaturated Fatty acids in heart failure patients. J Am Coll Cardiol. 2006 Oct 17;48(8):1600-6. doi: 10.1016/j.jacc.2006.05.073. Epub 2006 Sep 26. PMID 17045894
- [Background] Rusca A, Di Stefano AF, Doig MV, Scarsi C, Perucca E. Relative bioavailability and pharmacokinetics of two oral formulations of docosahexaenoic acid/eicosapentaenoic acid after multiple-dose administration in healthy volunteers. Eur J Clin Pharmacol. 2009 May;65(5):503-10. doi: 10.1007/s00228-008-0605-4. Epub 2009 Jan 16. PMID 19148629
- [Background] Raatz SK, Redmon JB, Wimmergren N, Donadio JV, Bibus DM. Enhanced absorption of n-3 fatty acids from emulsified compared with encapsulated fish oil. J Am Diet Assoc. 2009 Jun;109(6):1076-81. doi: 10.1016/j.jada.2009.03.006. PMID 19465191
- [Background] Skou HA, Toft E, Christensen JH, Hansen JB, Dyerberg J, Schmidt EB. N-3 fatty acids and cardiac function after myocardial infarction in Denmark. Int J Circumpolar Health. 2001 Aug;60(3):360-5. PMID 11590875
- [Background] Vidgren HM, Agren JJ, Schwab U, Rissanen T, Hanninen O, Uusitupa MI. Incorporation of n-3 fatty acids into plasma lipid fractions, and erythrocyte membranes and platelets during dietary supplementation with fish, fish oil, and docosahexaenoic acid-rich oil among healthy young men. Lipids. 1997 Jul;32(7):697-705. doi: 10.1007/s11745-997-0089-x. PMID 9252957
- [Background] Wang C, Harris WS, Chung M, Lichtenstein AH, Balk EM, Kupelnick B, Jordan HS, Lau J. n-3 Fatty acids from fish or fish-oil supplements, but not alpha-linolenic acid, benefit cardiovascular disease outcomes in primary- and secondary-prevention studies: a systematic review. Am J Clin Nutr. 2006 Jul;84(1):5-17. doi: 10.1093/ajcn/84.1.5. PMID 16825676